CLINICAL TRIAL: NCT02371967
Title: A Prospective Observational Study of Erivedge® Treatment, Effectiveness, and Safety Outcomes in Patients With Advanced Basal Cell Carcinoma
Brief Title: A Study to Assess the Effectiveness and Safety of Vismodegib (Erivedge®) in Participants With Advanced Basal Cell Carcinoma (BCC)
Acronym: ROSETT
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29507
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Basal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — HhAntag691

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- No Gorlin Syndrome Participants With No Prior HPI Exposure: BCC participants with advanced disease and no Gorlin syndrome, and who have not been exposed previously to an Hedgehog Pathway Inhibitor (HPI) (e.g., Vismodegib, LDE225) prior to diagnosis of advanced disease; will receive vismodegib therapy in compliance with the physician's standard practice as per local label and will be followed-up for approximately 3 years or until death, withdrawal of consent, sponsor's decision, lost to follow-up or end of study.
  Interventions: Drug: Vismodegib
- No Gorlin Syndrome Participants With Prior HPI Exposure: BCC participants with advanced disease and no Gorlin syndrome, and who have been exposed previously to an HPI (e.g., during clinical studies with vismodegib [SHH4476g {NCT00833417}, MO25616 {NCT01367665}] or LDE225); will receive vismodegib therapy in compliance with the physician's standard practice as per local label and will be followed-up for approximately 3 years or until death, withdrawal of consent, sponsor's decision, lost to follow-up or end of study.
  Interventions: Drug: Vismodegib
- Gorlin Syndrome Participants With/Without Prior HPI Exposure: BCC participants with advanced disease and Gorlin syndrome, and who have or have not been previously exposed to an HPI (e.g., during clinical studies); will receive vismodegib therapy in compliance with the physician's standard practice as per local label and will be followed-up for approximately 3 years or until death, withdrawal of consent, sponsor's decision, lost to follow-up or end of study.
  Interventions: Drug: Vismodegib

INTERVENTIONS:
Drug: Vismodegib — Vismodegib therapy will be given in compliance with the physician's standard practice as per local label.
  Other Names: Erivedge®

SUMMARY:
This prospective, observational, cohort study is designed to assess the effectiveness and safety outcomes of vismodegib and to assess actual day-to-day disease and participant management by the physician.

ELIGIBILITY:
Inclusion Criteria:

* BCC that meets one of the study's pre-specified cohort definitions
* Physician's decision to treat participant with vismodegib as per local label
* Participant who has not participated in a clinical trial within 90 days prior to study enrollment, with the exception of participants who meet the criteria for Cohort 2 (No Gorlin Syndrome Participants With Prior HPI Exposure)

Exclusion Criteria:

* Female participants are excluded if they are pregnant or if they plan to become pregnant during treatment or within 2 years after end of treatment
* Male participants with female partners of childbearing potential are excluded if they plan to impregnate their partner during treatment or within 2 months after end of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include adult participants with advanced BCC, in whom the treating physician has made the decision to commence vismodegib treatment (in accordance with the local label).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-04-08 (Actual); Primary Completion 2020-08-19 (Actual); Study Completion 2020-08-19 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Clinical Response as Assessed by Investigator According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1) | From the date of first treatment up to the date of progression or death from any cause (up to approximately 3 years)
Time to Clinical Response as Assessed by Investigator According to RECIST v1.1 | From the date of first treatment until the date of first documented confirmed complete response (CR) or partial response (PR) (whichever occurs first) (up to approximately 3 years)
Duration of Clinical Response as Assessed by Investigator According to RECIST v1.1 | From the date of occurrence of first clinical response up to the date of progression or death from any cause (up to approximately 3 years)
Percentage of Participants who Experience a Recurrence | From Baseline up to end of study (up to approximately 3 years)
Progression-Free Survival (PFS) as Assessed by Investigator According to RECIST v1.1 | From the date of first treatment up to the date of progression or death from any cause (up to approximately 3 years)
Overall survival (OS) | From the date of first treatment until death due to any cause (up to approximately 3 years)
Percentage of Participants With Adverse Events | From Baseline up to end of study (up to approximately 3 years)
Duration of Vismodegib Treatment | Baseline up to approximately 3 years
Percentage of Participants With Vismodegib Treatment Interruption | Baseline up to approximately 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- Sweden (4):
  - SU/Sahlgrenska, Hudkliniken, Gothenburg
  - Skånes Universitetssjukhus; Hudkliniken, Lund
  - Radiumhemmet, Solna
  - Norrlands universitetssjukhus; Onkologkliniken, Umeå